CLINICAL TRIAL: NCT00669331
Title: : A Phase III Multicenter, Randomized, Parallel Group, Controlled, Double Blind Study to Investigate the Safety and Efficacy of Inhaled Mannitol Over 12 Months in the Treatment of Bronchiectasis.
Brief Title: Inhaled Mannitol as a Mucoactive Therapy for Bronchiectasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Syntara (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DPM-B-305
Record Dates: First submitted 2008-04-28; First posted 2008-04-30 (Estimated); Results first posted 2016-04-29 (Estimated); Last update posted 2016-04-29 (Estimated); Status verified 2016-03

CONDITIONS: Bronchiectasis
Keywords: randomized clinical trial; mannitol; mucoactive
MeSH Terms: conditions — Bronchiectasis | interventions — Case-Control Studies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mannitol (Experimental): Inhaled mannitol 400mg
  Interventions: Drug: Inhaled mannitol
- Control (Placebo Comparator): Matched control - inhaled mannitol 50mg
  Interventions: Drug: Matched control

INTERVENTIONS:
Drug: Inhaled mannitol — 400mg dose of Mannitol BD (twice a day) for 52 weeks
  Arms: Mannitol
Drug: Matched control — 50mg dose of Mannitol BD (twice a day) for 52 weeks
  Arms: Control

SUMMARY:
No gold standard therapy exists for clearing mucus from the airways of patients with bronchiectasis. While rhDNase has a proven place in the treatment of cystic fibrosis (CF), it failed to improve Forced expiratory volume in one second (FEV1) in a short-term non-CF bronchiectasis study and has been shown to be detrimental after 6 months therapy in non CF bronchiectasis, moreover it has no proven effect on mucociliary clearance. Hypertonic saline has been shown to have a comparable mode of action to inhaled mannitol, but has yet to be examined as a long term treatment option in bronchiectasis.

The purpose of this study is to examine the efficacy and safety of 52 weeks treatment with inhaled mannitol in subjects with non-cystic fibrosis bronchiectasis. Previous studies with inhaled mannitol have demonstrated improvement in mucociliary clearance; mucus rehydration; improvement in quality of life and respiratory symptoms in patients with bronchiectasis and pulmonary function in cystic fibrosis. The results of this current study in combination with a recently completed 3 month study seek to confirm these early findings and to extend the evidence to support its use as a mucoactive therapy in subjects with bronchiectasis.

We hypothesize that mannitol will improve the overall health and hygiene of the lung through regular and effective clearing of the mucus load. As a consequence of the reduction in mucus load and inflammatory process, the frequency of bronchiectasis related pulmonary exacerbations and the need for exacerbation related antibiotic treatment should fall. Days in hospital and community health care costs are expected to change in line with improvements in respiratory health.

Finally, we plan to demonstrate that inhaled mannitol is safe and well tolerated over a 52 week period. We will test these hypotheses using 400 mg mannitol twice daily (BD) against control.

ELIGIBILITY:
Inclusion Criteria

1. Have given written informed consent to participate in this study in accordance with local regulations
2. Have documented evidence of confirmed diagnosis of (non-cystic fibrosis) bronchiectasis by computed tomography (CT), High resolution computed tomography (HRCT) or bronchogram
3. Be aged 18 - 85 years inclusive, male and female
4. Have FEV1 (Forced expiratory volume in one second) ≥ 40% and ≤85% predicted* and ≥1.0L (*according to NHANES III predicted tables) measured at Visit 0A (V0A)
5. Clinician documented history of at least 2 pulmonary exacerbations, each requiring antibiotic therapy, in the last 12 months prior to Visit 0A (V0A) and a total of at least 4 in the last 2 years prior to Visit 0A
6. Have a total SGRQ (St George's respiratory questionnaire) score of ≥30 at Visit 0B (V0B)
7. Have a production of ≥10g of sputum at Visit 0B Have reported chronic sputum production of ≥1 tablespoon (15mL) per day on the majority of days in the 3 months prior to Visit 0A
8. Be able to perform all the techniques necessary to measure lung function
9. Have FEV1 ≥40% predicted* and ≥1.0L (*according to NHANES III 1999 predicted tables) measured at V0B (Baseline result prior to MTT (Mannitol Tolerance Test) administration)

Exclusion Criteria

1. Be investigators, site personnel directly affiliated with this study, or their immediate families. Immediate family is defined as a spouse, parent, child or sibling, whether biologically or legally adopted.
2. Have bronchiectasis as a consequence of cystic fibrosis or focal endobronchial lesion or otherwise curable causes (e.g. foreign body aspiration)
3. Be considered "terminally ill" or listed for transplantation
4. Be using hypertonic saline in the 14 days prior to commencing Visit 0B or thereafter at any time during the study
5. Have previously used inhaled mannitol (Bronchitol) for more than a day
6. Have had a significant episode of hemoptysis (>60 mL) in the previous 6 months
7. Have had rescue antibiotics in the 4 weeks prior to V0B (chronic background antibiotic therapy accepted)
8. Have smoked within the last 3 months and must not smoke during their participation in the study
9. Have had a myocardial infarction in the three months prior to Visit 0A
10. Have had a cerebral vascular accident in the three months prior to Visit 0A
11. Have had major ocular surgery in the three months prior to Visit 0A
12. Have had major abdominal, chest or brain surgery in the three months prior to Visit 0A
13. Have a known cerebral, aortic or abdominal aneurysm
14. Have actively treated Mycobacterium tuberculosis
15. Have actively treated or unstable nontuberculous mycobacterial (NTM)infection or be under consideration for NTM treatment in the next 12 months
16. Have unstable Allergic bronchopulmonary aspergillosis (ABPA) requiring steroid therapy (≤5mg dose oral steroids in stable ABPA accepted)
17. Have end stage interstitial lung disease
18. Have active malignancy including melanoma (other skin carcinomas exempted). Remissions from any malignancy ≥2 years also exempted
19. Be breast feeding or pregnant, or plan to become pregnant while in the study
20. Be using an unreliable form of contraception (female subjects at risk of pregnancy only)
21. Be participating in another investigational drug study, parallel to, or within 4 weeks of Visit 0A
22. Have a known intolerance to mannitol or β2-agonists
23. Have uncontrolled hypertension - e.g. for adults: systolic blood pressure (BP) > 190 and or diastolic BP > 100
24. Subject has a condition or is in a situation which in the Investigator's opinion may put the subject at significant risk, may confound results or may interfere significantly with the patient's participation in the study
25. Have previously been screen failed for the study (exceptions - see section 3.3.2 Eligibility Criteria - Rescreening)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 485 (Actual)
Dates: Start 2009-11; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diana Bilton, MD, Principal Investigator — Brompton Hospital London UK; Greg Tino, MD, Principal Investigator — University of Pennsylvania Medical Centre, Philadelphia; Alan Barker, MD, Principal Investigator — Oregon Health Sciences University, Portland Oregon
Locations (83):
- United States (19):
  - National Jewish Medical and Research Center, Denver, Colorado
  - University of Connecticut Health Center, Pulmonary Division, Farmington, Connecticut
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - University of Miami, Miami, Florida
  - Florida Pulmonary Research, Winter Park, Florida
  - The University of Chicago Hospitals, Chicago, Illinois
  - Chest Medicine Clinical Services, LLC, Skokie, Illinois
  - Allergy and Critical Care Medicine Pulmonary Clinical Research Unit, Rochester, Minnesota
  - Saint Luke's Hospital, Chesterfield, Missouri
  - Pulmonary and Allergy Associates, Summit, New Jersey
  - Winthrop University Hospital, Mineola, New York
  - Research Associates of New York, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - The Oregon Clinic, PC/Pulmonary Division, Portland, Oregon
  - University of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - South Carolina Pharmaceutical Research, Spartanburg, South Carolina
  - Alamo Clinical Research Associates, San Antonio, Texas
  - Pulmonary Associates of Richmond, Inc, Richmond, Virginia
- Argentina (14):
  - Hospital Zonal Especializado en Agudos y Cronicos "Dr Antonio A. Cetrangolo, Florida Partido de Vicente López, Buenos Aires
  - Centro Respiratorio Quilmes, Quilmes, Buenos Aires
  - Instituto Argentino de Investigación Neurológica, Buenos Aires, Buenos Aires F.D.
  - Hospital Privado - Centro Medico de Cordoba, Córdoba, Córdoba Province
  - Insares, Mendoza, Mendoza Province
  - Centro Privado de Medicina Respiratoria, Entre Ríos, Paraná Entre Ríos
  - Hospital Interzonal General de Agudos "Dr Jose Penna", Bahia Bianca, Provinica de Buenos Aires
  - Corporacion medica de General San Martin, Matheu, San Martin Provincia de Buenos Aires
  - Clinica del Torax, Rosario, Santa Fe Province
  - Instituto Cardiovascular de Rosario, Rosario, Santa Fe Province
  - Sanatorio Parque, Rosario, Santa Fe Province
  - Investigaciones en Patologias Respiratorias, San Miguel de Tucumán, Tucumán Province
  - Centro Médico Dra. De Salvo, Buenos Aires
  - Atención Integral en Reumatología (AIR), Buenos Aires
- Australia (10):
  - Woolcock Institute of Medical Research, Glebe, New South Wales
  - St George Hospital, Kogarah, New South Wales
  - The Prince Charles Hospital, Chermside, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Repatriation General Hospital, Daws Park, South Australia
  - The Queen Elizabeth Hospital, Woodville, South Australia
  - St Vincent's Hospital, Fitzroy, Victoria
  - Western Hospital, Footscray, Victoria
  - The Rooms of Dr C Steinfort, Geelong, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria
- Belgium (3):
  - ULB Hopital Erasme - Department of Pneumology, Brussels, Brussels Capital
  - Cliniques Universitaires St. Luc (UCL) - Department of Pulmonology, Brussels, Brussels Capital
  - UZ Leuven (University Hospital Leuven) - Depatment of Pulmonary Medicine, Leuven, Leuven
- Chile (3):
  - Pontificia Universidad Catolica de Chile, Santiago, Santiago Metropolitan
  - Universidad de Chile, Santiago, Santiago Metropolitan
  - Hospital Regional de Talca, Talca, Talca
- Germany (4):
  - IKF Pneumologie GmbH and Co KG, Frankfurt am Main, Hesse
  - Medizinische Hochschule Hannover Klinik für Pneumologie, Hanover, Lower Saxony
  - Lungen und Bronchialheikunde, Bonn, North Rhine-Westphalia
  - Pneumologisch Studienzentrum, Leipzig, Saxony
- Netherlands (3):
  - Medisch Centrum Alkmaar - Department of Pulmonary Medicine, Alkmaar, Alkmaar AM
  - Atrium MC -Department of Pulmonary Diseases, Heerlen, Heerlen
  - Medisch Centrum Leeuwarden (MCL) - Department of Pulmonology, Leeuwarden, Leeuwarden AD
- New Zealand (3):
  - Middlemore Hospital, Auckland, Auckland
  - Green Lane Clinical Centre, Greenlane, Auckland
  - Waikato Hospital, Hamilton
- United Kingdom (24):
  - West Wales General Hospital, Carmarthen, Carmarthenshire
  - Royal Derby Hospital, Derby, Derbyshire
  - Royal Devon and Exeter Hospital, Exeter, Devon
  - Torbay Hospital, Torquay, Devon
  - Castle Hill Hospital, Cottingham, East Yorkshire
  - Glenfield Hospital, Leicester, Leicestershire
  - Nottingham City Hospital, Nottingham, Nottinghamshire
  - Churchill Hospital, Headington, Oxfordshire
  - Royal Shrewsbury Hospital, Shrewsbury, Shropshire
  - Sheffield Northern General Hospital, Sheffield, South Yorkshire
  - Stafford Hospital, Stafford, Staffordshire
  - Ashford & St Peters Hospital, Chertsey, Surrey
  - University Hospital of North Tees, Stockton, Teeside
  - Llandough Hospital, Cardiff, Vale of Glamorgan
  - Birmingam Queen Elizabeth Hospital, Birmingham, West Midlands
  - Wolverhampton New Cross Hospital, Wolverhampton, West Midlands
  - Aberdeen Royal Infirmary, Aberdeen
  - Belfast City Hospital, Belfast
  - University Hospital Aintree, Liverpool
  - Royal Brompton Hospital, London
  - Freeman Hospital, Newcastle upon Tyne
  - North Tyneside General Hospital, North Shields
  - Southampton General Hospital, Southampton
  - Wrexham Maelor Hospital, Wrexham

REFERENCES:
- [Background] Daviskas E, Anderson SD, Eberl S, Chan HK, Bautovich G. Inhalation of dry powder mannitol improves clearance of mucus in patients with bronchiectasis. Am J Respir Crit Care Med. 1999 Jun;159(6):1843-8. doi: 10.1164/ajrccm.159.6.9809074. PMID 10351929
- [Background] Daviskas E, Anderson SD, Eberl S, Young IH. Effect of increasing doses of mannitol on mucus clearance in patients with bronchiectasis. Eur Respir J. 2008 Apr;31(4):765-72. doi: 10.1183/09031936.00119707. Epub 2007 Dec 5. PMID 18057051
- [Background] Daviskas E, Anderson SD, Young IH. Inhaled mannitol changes the sputum properties in asthmatics with mucus hypersecretion. Respirology. 2007 Sep;12(5):683-91. doi: 10.1111/j.1440-1843.2007.01107.x. PMID 17875056
- [Background] Daviskas E, Anderson SD. Hyperosmolar agents and clearance of mucus in the diseased airway. J Aerosol Med. 2006 Spring;19(1):100-9. doi: 10.1089/jam.2006.19.100. PMID 16551221
- [Background] Daviskas E, Anderson SD, Gomes K, Briffa P, Cochrane B, Chan HK, Young IH, Rubin BK. Inhaled mannitol for the treatment of mucociliary dysfunction in patients with bronchiectasis: effect on lung function, health status and sputum. Respirology. 2005 Jan;10(1):46-56. doi: 10.1111/j.1440-1843.2005.00659.x. PMID 15691238
- [Background] Daviskas E, Robinson M, Anderson SD, Bye PT. Osmotic stimuli increase clearance of mucus in patients with mucociliary dysfunction. J Aerosol Med. 2002 Fall;15(3):331-41. doi: 10.1089/089426802760292681. PMID 12396422
- [Background] Daviskas E, Anderson SD, Eberl S, Chan HK, Young IH. The 24-h effect of mannitol on the clearance of mucus in patients with bronchiectasis. Chest. 2001 Feb;119(2):414-21. doi: 10.1378/chest.119.2.414. PMID 11171717
- [Derived] Bilton D, Tino G, Barker AF, Chambers DC, De Soyza A, Dupont LJ, O'Dochartaigh C, van Haren EH, Vidal LO, Welte T, Fox HG, Wu J, Charlton B; B-305 Study Investigators. Inhaled mannitol for non-cystic fibrosis bronchiectasis: a randomised, controlled trial. Thorax. 2014 Dec;69(12):1073-9. doi: 10.1136/thoraxjnl-2014-205587. Epub 2014 Sep 21. PMID 25246664

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Prior to randomisation, subjects underwent a Mannitol Tolerance Test (MTT) - only those who passed the MTT were eligible to be randomised. 581 patients in total underwent the MTT
Groups:
- Mannitol: Inhaled mannitol
  Inhaled mannitol: 400mg BD for 52 weeks
- Control: Matched control: Inhaled mannitol 50mg BD for 52 weeks
Period: Randomisation to First Dose
Arm/Group | Mannitol | Control
Started | 244 | 241
Completed | 233 | 228
Not Completed | 11 | 13
Not completed — Adverse Event | 1 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Lost to Follow-up | 2 | 0
Not completed — Death | 1 | 0
Not completed — Sponsor decision | 0 | 1
Not completed — Randomised in error | 3 | 10
Period: Blinded Treatment Period
Arm/Group | Mannitol | Control
Started | 233 | 228
Completed | 191 | 189
Not Completed | 42 | 39
Not completed — Adverse Event | 16 | 10
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 17 | 19
Not completed — Lost to Follow-up | 3 | 2
Not completed — Death | 0 | 2
Not completed — Physician Decision | 3 | 3
Not completed — Unable/unwilling to comply w trial reqs | 2 | 2

BASELINE CHARACTERISTICS:
Population: Patients randomised and treated with at least one dose of study medication
Groups:
- Total: Total of all reporting groups
Arm/Group | Mannitol | Control | Total
Number analyzed (Participants) | 233 | 228 | 461
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.30 (14.06) | 60.26 (13.02) | 59.77 (13.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 147 | 142 | 289
  Male | 86 | 86 | 172
Baseline Pulmonary Exacerbation rate [Mean (Standard Deviation); unit: events/year] | 3.20 (1.38) | 3.25 (1.40) | 3.22 (1.39)
Baseline % of Predicted FEV1 [Number; unit: participants]
  <60% | 101 | 107 | 208
  >=60% | 132 | 121 | 253
Extent of Bronchiectasis [Number; unit: participants]
  Diffuse | 133 | 118 | 251
  Focal | 77 | 73 | 150
  Both (Diffuse and Focal) | 23 | 37 | 60

OUTCOME MEASURES:

1. Primary Outcome: Rate of Graded Pulmonary Exacerbations
Description: A graded pulmonary exacerbation was defined as a worsening in signs and symptoms requiring a change in treatment (Center for Drug Evaluation and Research (CDER), 2007). Grade I was required 3 main signs and symptoms, Grade II 2 main signs and symptoms and Grade III 1 main and one or more minor signs and symptoms. Main signs and symptoms were increased cough, sputum volume or sputum purulence. Minor were upper respiratory tract infection, fever, increased wheezing, increased dyspnea, increase in respiratory rate, increase in cardiac frequency of >20%, and increased malaise, fatigue or lethargy. Rate is defined as the number of all GPE events observed in one treatment year
Time Frame: 52 weeks
Population: Randomised and Treated (referred to as the ITT population in this trial)
Measure: Number; unit: GPE events per year
Arm/Group | Mannitol | Control
Number analyzed (Participants) | 233 | 228
GPE events per year
  Raw rate | 1.95 | 2.10
  Rate from negative binomial model | 1.69 | 1.84
Statistical Analysis 1: Comparison: Mannitol vs Control; Test type: Superiority or Other; p = 0.3115, Negative binomial regression model; Negative binomial regression model with treatment, region and baseline PE rate as predictors and log of follow-up time as an offset variable; Rate Ratio Mannitol:Control = 0.92, 95% CI 2-sided [0.78 to 1.08] — For rate ratio, Mannitol rate is the numerator, Control rate is the denominator

2. Secondary Outcome: Quality of Life as Measured by the St. Georges Respiratory Questionnaire (SGRQ) Total Score
Description: The SGRQ was collected at baseline, week 6, week 16, week 28, week 40 and week 52. Change in total score was calculated from baseline. Total scores are a weighted sum across all questions. Scores are expressed as a percentage of overall impairment where 100 represents worst possible health status and 0 indicates best possible health status. Higher scores indicate lower quality of life. Outcome data table gives the raw mean total score at each visit.
Time Frame: 52 weeks
Population: Randomised and treated with one or more post-baseline SGRQ data available
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mannitol | Control
Number analyzed (Participants) | 228 | 219
units on a scale
  Baseline | 52.98 (14.64) | 52.22 (14.71)
  Week 6 | 44.09 (17.49) | 44.55 (18.49)
  Week 16 | 40.67 (19.07) | 44.23 (19.89)
  Week 28 | 41.45 (18.58) | 43.46 (19.05)
  Week 40 | 40.39 (18.86) | 43.51 (19.96)
  Week 52 | 41.43 (19.60) | 42.25 (19.50)
Statistical Analysis 1: Comparison: Mannitol vs Control; Test type: Superiority or Other; p = 0.0457, Mixed model repeated measures analysis; Model included treatment, visit, treatment*visit, region and baseline SGRQ Total score; LS mean difference across the 52 weeks = -2.40, 95% CI 2-sided [-4.76 to -0.05] — difference calculated Mannitol-control. Negative difference is in favour of mannitol since lower scores indicate improved quality of life

3. Secondary Outcome: Antibiotic Use Prescribed for Treated Pulmonary Exacerbations
Description: Rate of antibiotic treated graded pulmonary exacerbations, using the same definition of a graded pulmonary exacerbation as the primary endpoint. A graded pulmonary exacerbation was considered to be anti-biotic treated if use of oral, IV or inhaled antibiotic use was recorded related to the GPE event.
Time Frame: 52 weeks
Population: Randomised and treated (referred to as ITT)
Measure: Number; unit: events/year
Arm/Group | Mannitol | Control
Number analyzed (Participants) | 233 | 228
events/year | 1.9 | 2.1
Statistical Analysis 1: Comparison: Mannitol vs Control; Test type: Superiority or Other; p = 0.2754, Negative binomial regression model; Negative binomial regression model with treatment, region and baseline pulmonary exacerbation rate as predictors, log follow-up as offset; Rate ratio = 0.91, 95% CI 2-sided [0.77 to 1.08] — Rate ratio is for mannitol vs control

4. Secondary Outcome: Time to First Graded Exacerbation
Description: Time to first graded exacerbation is defined as the duration (in months) from the randomisation date to the start of the first reported graded PE during the on-treatment period. Patients without reported graded PE event will be censored at the last participation.
Time Frame: 52 weeks
Population: Randomised and treated
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Mannitol | Control
Number analyzed (Participants) | 233 | 228
months | 5.4 [4.1 to 6.7] | 4.1 [3.5 to 4.7]
Statistical Analysis 1: Comparison: Mannitol vs Control; Test type: Superiority or Other; p = 0.0218, Regression, Cox; Cox regression model was stratified by region and baseline PE rate; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.63 to 0.96]

5. Secondary Outcome: Duration of Graded Exacerbations
Description: Duration of graded exacerbations is defined as the number of days with graded PE within one treatment year. Mean days estimated via negative binomial model with treatment, region and baseline pulmonary exacerbation rate as predictors, with log of follow-up time as the offset variable
Time Frame: 52 weeks
Population: Randomised and treated
Measure: Mean (95% Confidence Interval); unit: Days with GPE
Arm/Group | Mannitol | Control
Number analyzed (Participants) | 233 | 228
Days with GPE | 31.49 [25.54 to 38.82] | 35.74 [28.90 to 44.20]
Statistical Analysis 1: Comparison: Mannitol vs Control; Analysed using a negative binomial model with treatment, region and baseline pulmonary exacerbation rate as predictors, and with log of follow-up time as the offset variable; Test type: Superiority or Other; p = 0.3602, Negative binomial model; treatment, region and baseline pulmonary exacerbation rate as predictors, and with log of follow-up time as the offset variable; Rate ratio = 0.88, 95% CI 2-sided [0.67 to 1.16]

6. Secondary Outcome: Sputum Volume
Description: 24 hour sputum weight, measured at baseline, week 6, week 16, week 28, week 40, week 52
Time Frame: 52 weeks
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Mannitol | Control
Number analyzed (Participants) | 233 | 228
g
  Baseline | 28.88 (18.71) | 28.96 (19.92)
  Week 6 | 24.97 (23.17) | 22.82 (20.06)
  Week 16 | 23.69 (22.09) | 20.25 (16.99)
  Week 28 | 22.92 (25.66) | 18.88 (17.83)
  Week 40 | 21.56 (21.58) | 18.17 (16.67)
  Week 52 | 20.54 (24.07) | 18.33 (16.00)
Statistical Analysis 1: Comparison: Mannitol vs Control; Test type: Superiority or Other; p = 0.0355, Mixed Models Analysis; Model includes treatment, visit, treatment*visit, region and baseline sputum weight (g); ls mean difference across 52 weeks = 2.76, 95% CI 2-sided [0.19 to 5.33] — Difference mannitol-control

7. Secondary Outcome: Daytime Sleepiness Scores
Description: Epworth Sleepiness Scale (ESS) score was calculated as the sum of scores for each of eight individual questions, such that a total score of zero represents no daytime sleepiness, and a total score of 24 represents the maximum degree of daytime sleepiness. Measured at baseline, 6 weeks, 16 weeks, 28 weeks, 40 weeks, 52 weeks
Time Frame: 52 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mannitol | Control
Number analyzed (Participants) | 233 | 228
units on a scale
  Baseline | 7.23 (4.85) | 6.89 (4.89)
  Week 6 | 6.07 (4.78) | 6.87 (4.74)
  Week 16 | 6.21 (5.10) | 6.50 (4.86)
  Week 28 | 6.05 (4.73) | 6.57 (4.82)
  Week 40 | 6.32 (5.10) | 6.33 (4.83)
  Week 52 | 6.09 (4.98) | 6.34 (5.02)
Statistical Analysis 1: Comparison: Mannitol vs Control; Test type: Superiority or Other; p = 0.1159, Mixed Models Analysis; Model includes treatment, visit, treatment*visit, region and baseline ESS score; LS mean diff across post-baseline visits = -0.44, 95% CI 2-sided [-0.99 to 0.11] — Negative change indicates an improvement in ESS score. Difference calculated Mannitol - Control

8. Secondary Outcome: Lung Function - Change in FEV1 (Forced Expiratory Volume in One Second)
Time Frame: 52 weeks
Population: Randomised and treated with at least one post-baseline spirometry assessment
Measure: Least Squares Mean (95% Confidence Interval); unit: mL
Arm/Group | Mannitol | Control
Number analyzed (Participants) | 229 | 219
mL | 2.36 [-24.03 to 28.74] | -5.20 [-32.35 to 21.95]
Statistical Analysis 1: Comparison: Mannitol vs Control; Test type: Superiority or Other; p = 0.6677, Mixed Models Analysis; Model of absolute change from baseline in FEV1. Model includes terms for treatment, visit, trt*visit, region and baseline value; Mean Difference (Net) = 7.56, 95% CI 2-sided [-27.01 to 42.13] — ls mean difference Mannitol-Control

9. Secondary Outcome: Lung Function - Change in FVC (Forced Vital Capacity)
Time Frame: 52 weeks
Population: Randomised and treated with at least one post-baseline spirometry assessment
Measure: Least Squares Mean (95% Confidence Interval); unit: mL
Arm/Group | Mannitol | Control
Number analyzed (Participants) | 229 | 219
mL | 0.15 [-36.75 to 37.05] | -15.70 [-53.64 to 22.25]

10. Secondary Outcome: Lung Function - Change in FEV1/FVC
Description: FEV1 expressed as a ratio of FVC. Endpoint is expressed as a percentage ie FEV1/FVC*100
Time Frame: 52 weeks
Population: Randomised and treated with at least one post-baseline spirometry assessment
Measure: Least Squares Mean (95% Confidence Interval); unit: ratio (expressed as a %)
Arm/Group | Mannitol | Control
Number analyzed (Participants) | 229 | 219
ratio (expressed as a %) | -0.08 [-0.68 to 0.53] | 0.09 [-0.52 to 0.71]

11. Secondary Outcome: Lung Function - Change in FEF25-75 (Forced Expiratory Flow Rate Averaged Over 25th -75th Percentile of FVC)
Time Frame: 52 weeks
Population: Randomised and treated with at least one post-baseline spirometry assessment
Measure: Least Squares Mean (95% Confidence Interval); unit: mL/s
Arm/Group | Mannitol | Control
Number analyzed (Participants) | 229 | 219
mL/s | -18.21 [-59.09 to 22.67] | -3.40 [-45.28 to 38.47]

12. Secondary Outcome: Safety Profile - Sputum Microbiology
Description: sputum microbiology assessed as the presence of abnormal flora in sputum sample taken at any post baseline visit
Time Frame: 52 weeks
Measure: Number; unit: participants
Arm/Group | Mannitol | Control
Number analyzed (Participants) | 233 | 228
participants | 81 | 81

13. Secondary Outcome: Safety Profile - Clinical Chemistry
Description: Clinical chemistry was assessed as clinically significant abnormal liver function test and clinically significant abnormal urea/electrolyte test at any point post baseline.
Time Frame: 52 weeks
Measure: Number; unit: participants
Arm/Group | Mannitol | Control
Number analyzed (Participants) | 233 | 288
participants
  Subjects with Clin sig liver funtion tests at wk52 | 2 | 0
  Subjects with clin sig urea/electrolyte test wk52 | 3 | 0

14. Secondary Outcome: Safety Profile - Hematology
Description: hematology assessed as clinically significant abnormal FBC (Full Blood count) at any point post baseline.
Time Frame: 52 weeks
Measure: Number; unit: participants
Arm/Group | Mannitol | Control
Number analyzed (Participants) | 233 | 228
participants | 13 | 5

15. Secondary Outcome: • (Exploratory) Number of Hospitalizations Due to Pulmonary Exacerbations
Description: Mean rate of hospitalisations (number/year) summarised and analysed to take account of differing follow-up times.
Time Frame: 52 weeks
Measure: Mean (95% Confidence Interval); unit: hospitalisations/year
Arm/Group | Mannitol | Control
Number analyzed (Participants) | 233 | 228
hospitalisations/year | 0.12 [0.07 to 0.20] | 0.20 [0.13 to 0.31]
Statistical Analysis 1: Comparison: Mannitol vs Control; Test type: Superiority or Other; p = 0.0928, Negative binomial regression; Rate ratio = 0.61, 95% CI 2-sided [0.34 to 1.09]

16. Other Pre Specified Outcome: Health Related Costs of Treating Patients With Bronchiectasis
Description: In the presence of a significant primary endpoint, these data were intended to be derived using the trial data together with external information (Note as the primary objective of this study did not reach statistical significance, health related costs were not assessed)
Time Frame: 52 weeks
Population: No data were collected. Since the primary objective was not significant in this study, further exploration of health economic endpoints was not done.
Groups:
- Mannitol: Inhaled mannitol 400mg
  Inhaled mannitol: 400mg dose of Mannitol BD for 52 weeks
- Control: Matched control - inhaled mannitol 50mg
  Matched control: 50mg dose of Mannitol BD for 52 weeks
Arm/Group | Mannitol | Control
Number analyzed (Participants) | 0 | 0

17. Other Pre Specified Outcome: Health Status and Utility Scores
Description: In the presence of a significant primary endpoint, these data were intended to be derived from the trial data and external information (Note as the primary objective of this study did not reach statistical significance, differences in health status and utility scores were not assessed)
Time Frame: 52 weeks
Population: No data were collected. As the primary objective of this study did not reach statistical significance, health status and utility scores were not derived.
Arm/Group | Mannitol | Control
Number analyzed (Participants) | 0 | 0

18. Other Pre Specified Outcome: Health Related Quality of Life (HRQL) and Quality Adjusted Life Years (QALYs) by Treatment Group Using Utility Scores From the Health Utilities Index Questionnaire
Description: In the presence of a significant primary endpoint, these data were intended to be derived using the trial data and external information (Note as the primary objective of this study did not reach statistical significance, HRQL and QALYs were not collected).
Time Frame: 52 weeks
Population: No data were collected for this assessment. As the primary objective of this study did not reach statistical significance, HRQL and QALYs were not derived.
Arm/Group | Mannitol | Control
Number analyzed (Participants) | 0 | 0

19. Other Pre Specified Outcome: Cost Effectiveness of Treating Patients With Bronchiectasis With Inhaled Mannitol
Description: In the presence of a significant primary endpoint, these data were intended to be derived using the trial data and external information (Note as the primary objective of this study did not reach statistical significance, cost effectiveness was not collected).
Time Frame: 52 weeks
Population: Not collected. As the primary objective of this study did not reach statistical significance, cost effectiveness data were not collected.
Arm/Group | Mannitol | Control
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 52 weeks
Arm/Group | Mannitol | Control
Serious Adverse Events (participants affected / at risk) | 43/233 | 51/228
Other Adverse Events (participants affected / at risk) | 215/233 | 214/228
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mannitol (N=233) | Control (N=228)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Angina Pectoris (Cardiac disorders) | 1 | 0
Cardiac Failure Congestive (Cardiac disorders) | 1 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 2
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 1
Catheter related complication (General disorders) | 1 | 0
Chest pain (General disorders) | 2 | 0
Condition Aggravated (General disorders) | 21 | 26
Disease prodomal stage (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 0 | 1
Cholecystisis (Hepatobiliary disorders) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
Dacryocystisis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Lobar pneumonia (Infections and infestations) | 1 | 2
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Lung abscess (Infections and infestations) | 1 | 0
Lung infection pseudomonal (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 7 | 7
Swine Influenza (Infections and infestations) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Fibula Fracture (Injury, poisoning and procedural complications) | 1 | 0
Seroma (Injury, poisoning and procedural complications) | 0 | 1
Skin lacreation (Injury, poisoning and procedural complications) | 2 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Transient global amnesia (Nervous system disorders) | 0 | 1
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1 | 0
Varicocele (Reproductive system and breast disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pharyngeal pouch (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bladder repair (Surgical and medical procedures) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mannitol (N=233) | Control (N=228)
Diarrhoea (Gastrointestinal disorders) | 15 | 21
Nausea (Gastrointestinal disorders) | 14 | 18
Condition aggravated (General disorders) | 149 | 159 — INCLUDES SERIOUS ADVERSE EVENTS ALSO
Lower respiratory tract infection (Infections and infestations) | 16 | 21 — INCLUDES SERIOUS ADVERSE EVENTS ALSO
Lower respiratory tract infection bacterial (Infections and infestations) | 12 | 9
Nasopharyngitis (Infections and infestations) | 36 | 30
Sinusitis (Infections and infestations) | 17 | 14
Bacteia sputum identified (Investigations) | 30 | 30
Back pain (Musculoskeletal and connective tissue disorders) | 19 | 13
Headache (Nervous system disorders) | 27 | 32
Cough (Respiratory, thoracic and mediastinal disorders) | 30 | 22
Dsypnoea (Respiratory, thoracic and mediastinal disorders) | 20 | 16 — INCLUDES SERIOUS ADVERSE EVENTS ALSO
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 24 | 23 — INCLUDES SERIOUS ADVERSE EVENTS ALSO
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 | 18

LIMITATIONS AND CAVEATS:
Relatively few studies in this area -ideal choice of endpoints not well-defined. No widely accepted exacerbation definition. Relies on patients' accurate & timely symptom reporting.Unclear event end-dates may impact on counting of subsequent events.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less